CLINICAL TRIAL: NCT00000378
Title: Antidepressant Treatment of Melancholia in Late :Ife
Brief Title: Antidepressant Treatment of Melancholia in Late Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #3105; R01MH055716 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2008-09

CONDITIONS: Depression; Melancholia
Keywords: Aged; Antidepressive Agents, Tricyclic; Depression; Female; Human; Male; Middle Age; Nortriptyline; Sertraline; Serotonin Uptake Inhibitors; Antidepressive Agents, Tricyclic -- *therapeutic use; Antidepressive Agents, Tricyclic -- adverse effects; Depression -- *drug therapy; Nortriptyline -- *therapeutic use; Nortriptyline -- adverse effects; Sertraline -- *therapeutic use; Sertraline -- adverse effects; Serotonin Uptake Inhibitors -- *therapeutic use; Serotonin Uptake Inhibitors -- adverse effects
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Sertraline; Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sertaline (Active Comparator): patients randomized to sertraline 12 week trial does up to 200mgs
  Interventions: Drug: Sertraline
- nortriptyline (Active Comparator): patients randomized to nortriptyline dose adjusted to therapeutic level
  Interventions: Drug: Nortriptyline

INTERVENTIONS:
Drug: Sertraline — 12 week trial dose up to 200mgs
  Arms: sertaline
Drug: Nortriptyline — 12 week trial dose adjusted to therapeutic level
  Other Names: nortiptyline
  Arms: nortriptyline

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of a select serotonin re-uptake inhibitor (SSRI, sertraline) and a tricyclic antidepressant (TCA, nortriptyline) in outpatients over the age of 60 who have major depression.

SSRIs are effective in the treatment of major depression. However, there is also evidence that SSRIs may be significantly less effective than TCAs for patients with late-life major depression with melancholia. Since SSRIs seem to be easier to take than TCAs and are more widely prescribed, it is important to determine which of these types of antidepressants works best to treat these patients.

Patients will be assigned randomly to receive either sertraline (a SSRI) or nortriptyline (a TCA) for 12 weeks. Patients will be monitored for symptoms, side effects, and quality of life. If a patient responds to treatment, he/she will participate in a 6-month continuation phase in which he/she will continue to receive the same medication.

An individual may be eligible for this study if he/she:

Has unipolar major depression (with some exceptions) and is over 60 years old.

DETAILED DESCRIPTION:
To compare the efficacy and safety of a select serotonin re-uptake inhibitor (SSRI, sertraline) and a tricyclic antidepressant (TCA, nortriptyline) in outpatients over the age of 60 who meet Diagnostic and Statistical Manuel-IV criteria for unipolar major depression, excluding patients who meet criteria for psychotic or atypical subtype. To test the hypothesis that medication condition interacts with diagnostic subtype (melancholic vs non-melancholic) in determining antidepressant response. To examine the roles of symptom severity and alternative diagnostic subtyping in contributing to this pattern.

SSRIs are effective in the treatment of major depression. However, there is also evidence that SSRIs may be significantly less effective than TCAs for depressed patients with melancholia. This issue is of particular concern in late-life major depression. SSRIs have important safety advantages with respect to overdose and a benign cardiovascular profile. Furthermore, the SSRIs do not have significant anticholinergic effects, and appear to be better tolerated than the TCAs. Perhaps most important, the SSRIs currently are prescribed widely as the medication treatment of first choice for major depression in late life. Therefore, if it were determined that SSRIs are considerably less effective than TCAs in the treatment of melancholia in the elderly, there would be significant ramifications for clinical practice.

Randomization to sertraline (a SSRI) or nortriptyline (a TCA) is stratified by the presence or absence of melancholia. Outcome measures for the 12-week acute phase include clinician and patient ratings of symptoms, side effects, and an evaluation of the health-related quality of life (HRQOL). At the end of the acute treatment phase, patients who meet criteria for clinical response participate in a 6-month continuation phase.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Unipolar major depression (per Diagnostic and Statistical Manuel-IV criteria) with or without melancholia.

Exclusion Criteria:

-

Patients with the following symptoms or conditions are excluded:

Psychotic or atypical subtype of unipolar major depression.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 1997-07; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Roose, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- 1051 Riverside Drive, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sertaline | Nortriptyline
Started | 58 | 52
Completed | 42 | 38
Not Completed | 16 | 14
Not completed — Lack of Efficacy | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertaline | Nortriptyline | Total
Number analyzed (Participants) | 58 | 52 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 50 | 48 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 58 | 52 | 110

OUTCOME MEASURES:

1. Primary Outcome: HAMILTON Rating Scale for DEPRESSION Range
Description: Hamilton scale range 0-40, values below 7 are considered normal. the higher the number the more severe the depression weekly assessments, The primary outcome is a comparison of the baseline Hamilton to the 12 week measurement
Time Frame: BASELINE COMPARED TO 12 WEEK MEASUREMENT
Population: intent to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertaline | Nortriptyline
Number analyzed (Participants) | 58 | 52
units on a scale
  BASELINE | 27.3 (6.6) | 27.1 (4.4)
  12 WEEK DATA | 10.7 (8.3) | 8.4 (7.7)
Statistical Analysis 1: Comparison: Sertaline vs Nortriptyline; logistic regression and mixed effects model; Test type: Superiority or Other; p < 0.05, Regression, Logistic — actual calculation

ADVERSE EVENTS:
Arm/Group | Sertaline | Nortriptyline
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/52
Other Adverse Events (participants affected / at risk) | 2/58 | 4/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sertaline (N=58) | Nortriptyline (N=52)
orthostatic hypotension (Cardiac disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No